CLINICAL TRIAL: NCT00153530
Title: Phase IV Study on the Role of Whole Brain Irradiation in Primary CNS Lymphoma (PCNSL) After High-dose Methotrexate
Brief Title: Whole Brain Irradiation in Primary Central Nervous System (CNS) Lymphoma (PCNSL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Agnieszka Korfel, G-PCNSL-SG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-PCNSL-SG1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-07

CONDITIONS: Central Nervous System Lymphoma
Keywords: primary central nervous system lymphoma
MeSH Terms: interventions — Methotrexate; Radiotherapy

ARMS (2):
- 1 (Active Comparator): 1 chemotherapy with radiotherapy
  Interventions: Drug: methotrexate; Radiation: radiotherapy
- 2 (Experimental): chemotherapy without radiotherapy
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: methotrexate — 1. chemotherapy with radiotherapy
  2. chemotherapy without radiotherapy
Radiation: radiotherapy — whole-brain irradiation
  Arms: 1

SUMMARY:
The aim of the study is to deliver primary systemic high-dose methotrexate (MTX) treatment to PCNSL patients and to define the role of whole brain irradiation (WBI) in primary therapy, i.e., to analyze whether patients who have undergone primary chemotherapy can postpone irradiation with its possible late sequelae until recurrence without incurring losses in progression-free and overall survival. This is studied here for the first time worldwide in a systematic, controlled and randomized manner. In this study, one arm with six cycles of high-dose MTX and subsequent irradiation (A1), which comes closest to a "standard arm of primary therapy", at least according to the majority assessment, is compared to irradiation at recurrence with regard to time to progression and overall survival (A2). In primary therapy failure, it will also be analyzed to what extent salvage therapy with AraC is equivalent to irradiation as the "standard arm" with regard to time to progression and overall survival (arm B1 and B2).

DETAILED DESCRIPTION:
Six 14-day cycles of high-dose MTX will be given at the beginning of the study. Randomization will be performed centrally at the study headquarters in UKBF Berlin already at study inclusion. Patients meeting all inclusion criteria will receive the first systemic treatment with 4 g/m2 MTX i.v. over 4 hours within 14 days. Dexamethasone in a dose of 3 x 8 mg/day orally for 10 days will additionally be given in the first cycle. This dexamethasone dose will be started 3 days before the first MTX application. Ten to 14 days after the 3rd and 6th MTX dose, the response to MTX therapy will be evaluated by MRI and a repeated CSF examination in the case of renewed CSF involvement. Assessment can also be made at any other time point if there is clinical deterioration. In all cases, the neuroradiological reference center (Department of Neuroradiology, University of Tübingen) will decide about the response to MTX therapy. MRI and CT scans should be sent to the neuroradiological reference center after HD MTX is terminated for central response evaluation. If complete remission is achieved after completing high-dose MTX therapy, patients will be treated with WBI (45 Gy in 1.5 Gy fractions) starting a minimum of 4 and a maximum of 7 weeks after the end of chemotherapy (arm A1) or WBI at first recurrence (arm A2). If primary therapy is not successful (partial remission, stable disease after the 6th cycle, progression at any time of MTX therapy), patients will receive WBI (45 Gy in 1.5 Gy fractions; arm B1) or high-dose AraC chemotherapy 3 g/m2 i.v. over 3 hours every 12 hours for 2 days (arm B2) according to the randomization. If high-dose MTX therapy leads to termination before the application of 6 cycles of MTX (see termination criteria) but allows further AraC therapy or WBI, further treatment is given in the non-CR arm according to the randomization. High-dose AraC therapy will be administered in four 3-week cycles. If complete remission occurs already after one or two cycles, only one additional cycle will be applied. Patients will not be crossed over into the B arms.

If there is a recurrence or progression after finishing a complete treatment arm, the patient can be treated with chemotherapy according to PCV protocol or WBI in the B2 arm. This decision is left up to the individual study center.

The G-PCNSL-SG-1 study is a prospective, controlled phase IV study with central randomization. Patients in both arms will be submitted to stratified randomization according to age (< 60; > 60) and center to minimize the effect of important therapy-related prognostic factors. The study is not blinded. Randomization will be performed centrally at study inclusion at the Institute of Medical Informatics, Biometry and Epidemiology, University Hospital Benjamin Franklin of the Free University of Berlin.

The planned study duration is 7 years - 4 years in the recruitment phase with a subsequent 3-year follow-up period and a 6-month evaluation phase. For an individual patient, the treatment time in arm A1 is 12 weeks for 6 cycles of MTX therapy, followed by a 4-7-week resting period and then 6 weeks until the completion of WBI (arm A1). In arm A2, the patient is irradiated (a total of 6 weeks) only in the case of recurrence. Up to that point, the patient will be followed up in fixed intervals like those patients in A1 after WBI. In arm B, MTX therapy is immediately followed by 6 weeks of WBI (arm B1) or the maximal 3 months of AraC therapy. After completing the protocol of the planned therapy, all patients will be followed-up for at least three years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically/immunocytologically confirmed primary non-Hodgkin's lymphoma of the CNS. A central reference pathological report will be made on inclusion into the study (Prof. Dr. Pietsch, Reference Center for Brain Tumors of the German Society for Neuropathology and Neuroanatomy, Institute of Neuropathology of the Bonn University Hospital). Histological diagnosis is usually performed by preferential stereotactic biopsy of suspicious lesions in the brain or spinal cord. The diagnosis from cerebrospinal fluid (CSF) requires the detection of malignant lymphocytes according to cytological and immunocytological criteria. There should be no more than 2 weeks between establishing the diagnosis and inclusion in the study. The availability of the reference pathological report is not absolutely necessary for inclusion in the study and beginning therapy.
* Aged > 18 years
* Life expectancy of at least 2 months
* Adequate bone marrow reserve with a peripheral granulocyte count of > 1,500/µl and thrombocyte count of > 100,000/µl; bilirubin in the normal range; GOT of < three times the upper normal limit and adequate renal function with a creatinine clearance of > 50 ml/min and serum creatinine in the normal range.
* Written informed consent
* In women of child-bearing age, pregnancy is excluded, effective contraception is necessary, and women should not be breast feeding.

Exclusion Criteria:

* Manifestation of lymphoma outside of the CNS
* Severe diseases in other organs which would make performing intensive chemotherapy impossible; Karnofsky index > 50% due to previous diseases other than PCNSL. Karnofsky > 30 will be accepted only due to the PCNSL.
* Active infection
* HIV positivity
* Previous treatment of PCNSL other than with corticosteroids, antiepileptics or diuretics
* Previous radiotherapy of the brain
* Concomitant or previous malignant diseases in the last 5 years except for an adequately treated basal cell carcinoma or cervical carcinoma in situ
* Immunosuppression, concomitant immunosuppressive therapy, or organ transplantation
* Ongoing chemotherapy for another disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Estimated)
Dates: Start 2000-05; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
progression-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Thiel, MD, Principal Investigator — Charite Campus Benjamin Franklin
Locations (1):
- Charite Campus Benjamin Franklin, Berlin, Germany

REFERENCES:
- [Derived] Thiel E, Korfel A, Martus P, Kanz L, Griesinger F, Rauch M, Roth A, Hertenstein B, von Toll T, Hundsberger T, Mergenthaler HG, Leithauser M, Birnbaum T, Fischer L, Jahnke K, Herrlinger U, Plasswilm L, Nagele T, Pietsch T, Bamberg M, Weller M. High-dose methotrexate with or without whole brain radiotherapy for primary CNS lymphoma (G-PCNSL-SG-1): a phase 3, randomised, non-inferiority trial. Lancet Oncol. 2010 Nov;11(11):1036-47. doi: 10.1016/S1470-2045(10)70229-1. Epub 2010 Oct 20. PMID 20970380
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/17301290?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=75